CLINICAL TRIAL: NCT07163585
Title: Safety and Efficacy of Oral Brivaracetam Versus Levetiracetam as Monotherapy in Children Aged 1 Month to 14 Years With Newly Diagnosed Epilepsy
Brief Title: Comparison of Oral Brivaracetam Versus Levetiracetam as Monotherapy in Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RESnTEC, Institute of Research (Other)
Responsible Party: Principal Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dr-Ikram-CH-Multan
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam; Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brivaracetam group (Experimental): Patients were given oral brivaracetam in a dose of 1-2 mg/kg/day in two divided doses, titrated to a maximum of 5 mg/kg/day based on clinical response and tolerability.
  Interventions: Drug: Brivaracetam
- Levetiracetam group (Experimental): Oral levetiracetam was initiated at a dose of 10-20 mg/kg/day in two divided doses, with gradual escalation up to 60 mg/kg/day if needed.
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Brivaracetam — Brivaracetam was initiated at a dose of 1-2 mg/kg/day in two divided doses, titrated to a maximum of 5 mg/kg/day based on clinical response and tolerability.
  Arms: Brivaracetam group
Drug: Levetiracetam — Levetiracetam was initiated at a dose of 10-20 mg/kg/day in two divided doses, with gradual escalation up to 60 mg/kg/day if needed.
  Arms: Levetiracetam group

SUMMARY:
Despite increasing clinical use of both agents, there is a paucity of head-to-head comparative data on the safety and efficacy of brivaracetam versus levetiracetam as initial monotherapy in children. The present study was therefore designed to compare the safety and efficacy of oral brivaracetam and levetiracetam as monotherapy in children aged one month to 14 years with newly diagnosed epilepsy.

DETAILED DESCRIPTION:
Most existing studies have focused on adjunctive use or refractory epilepsy, while evidence in treatment-naïve pediatric populations remains sparse. Addressing this gap is critical, as early and effective seizure control can substantially influence long-term neurodevelopmental outcomes. By evaluating seizure outcomes, tolerability, and adverse effect profiles, this study aims to provide evidence to guide clinicians in selecting the most appropriate first-line anti-seizure medication (ASM) for pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Children of either gender
* Aged 1 month to 14 years
* With a clinical diagnosis of newly diagnosed epilepsy

Exclusion Criteria:

* History of prior use of long-term antiseizure medications
* Evidence of progressive neurological disease
* Metabolic abnormalities
* Structural brain malformations
* Incompatible with monotherapy
* Severe systemic comorbidities

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Cessation of seizures | Up to 3 months
  Cessation of seizures was labeled "yes" when a patient remained seizure free.

SECONDARY OUTCOMES:
Adverse events | Up to 3 months
  Labeled "yes" if any treatment-related adverse events reported.

CONTACTS AND LOCATIONS:
Overall Officials: Ikram Rahman, Principal Investigator — Children's Hospital and institute of Child Health Multan, Pakistan; Nuzhat Rahman, FCPS, Study Director — Children's Hospital and institute of Child Health Multan, Pakistan
Locations (1):
- The Children's Hospital and Institute of Child Health, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.